CLINICAL TRIAL: NCT04494503
Title: A Phase Ib/II Study of the Safety, Pharmacokinetic, Pharmacodynamic and Efficacy of APG-2575 Single Agent and in Combination With Other Therapeutic Agents in Patients With Relapsed/Refractory CLL/SLL
Brief Title: Study of APG2575 Single Agent and Combination Therapy in Patients With Relapsed/Refractory CLL/SLL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG2575CC101
Record Dates: First submitted 2020-07-21; First posted 2020-07-31 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: APG-2575; rituximab; ibrutinib; chronic lymphocytic leukemia(CLL); small lymphocytic lymphoma(SLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lisaftoclax; Rituximab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- APG-2575 single agent in Relapse/Refractory CLL/SLL (Experimental): APG-2575 orally once daily at 400mg, 600mg, 800mg dose levels respectively, every 28 days as a cycle.
  Interventions: Drug: APG-2575
- APG-2575+Rituximab in Relapse/Refractory CLL/SLL (Experimental): Stage 1:APG-2575 orally once daily starting from 200mg and will be increased in subsequent cohorts to 400mg, 600mg, 800mg. Rituximab 375mg/m2 ivgtt on C1D8 and 500mg/m2 ivgtt on C2-6D1. Every 28 days as a cycle.
  Stage 2: APG-2575 MTD/RP2D combined with rituximab. Every 28 days as a cycle.
  Interventions: Drug: APG-2575; Drug: Rituximab
- APG-2575+ibrutinib in Relapse/Refractory CLL/SLL (Experimental): Stage 1: APG-2575 orally once daily starting from 200mg and will be increased in subsequent cohorts to 400mg, 600mg, 800mg.Ibrutinib 420mg orally once daily during C1D8-28 and following cycles. Every 28 days as a cycle.
  Stage 2: APG-2575 MTD/RP2D combined with ibrutinib. Every 28 days as a cycle.
  Interventions: Drug: APG-2575; Drug: Ibrutinib

INTERVENTIONS:
Drug: APG-2575 — APG-2575 orally once daily, every 28 days as a cycle.
Drug: Rituximab — Rituximab 375mg/m2 ivgtt on C1D8 and 500mg/m2 ivgtt on C2-6D1.
  Arms: APG-2575+Rituximab in Relapse/Refractory CLL/SLL
Drug: Ibrutinib — Ibrutinib 420mg orally once daily during C1D8-28 and following cycles.
  Arms: APG-2575+ibrutinib in Relapse/Refractory CLL/SLL

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetic, pharmacodynamic and efficacy of APG-2575 single agent and in combination with other therapeutic agents in patients with relapsed/refractory CLL/SLL.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase Ib/II study of safety, PK, PD and efficacy of APG-2575 as a single agent or in combination with rituximab or ibrutinib in relapsed/refractory CLL/SLL patients.

This study consists of two parts: The first part is the APG-2575 single agent cohort expansion. The cohort expansion will be conducted at three dose levels of 400 mg, 600 mg, and 800 mg. And up to 15 patients are planned to be enrolled at each dose level.

The second part contains two arms: APG-2575 combined with rituximab (Arm A) and APG-2575 combined with ibrutinib (Arm B). Both the two arms consist of two stages: dose escalation stage (first stage) and dose expansion stage (second stage). The first stage is the study of APG-2575 dose escalation combined with rituximab/ibrutinib. APG-2575 dose escalates according to the standard 3+3 design, the initial dose is 200mg, the dose of APG-2575 will be increased in subsequent levels, to 400mg, 600mg, 800mg respectively. The second stage is the MTD/RP2D expansion stage. Once the respective MTD/RP2D of arms A and B is determined, up to 15 subjects in each MTD/RP2D dose level would be enrolled.

APG-2575 will be administered orally, once daily for consecutive 4 weeks as one cycle.

Rituximab, on cycle 1 day 8(C1D8): 375mg/m2; on cycles 2-6 day l(C2-6D1): 500mg/m2, a total of six infusions.

Ibrutinib 420 mg will be orally administered daily beginning from cycle 1 day 8 and continuously thereafter, every 4 weeks as a cycle.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet each of the following inclusion criteria are eligible to participate in this study:

1. Age ≥18 years old.
2. Diagnosis as relapsed/refractory chronic lymphocytic leukemia/ small lymphocytic lymphoma according to the IWCLL NCI-WG guidelines revised in 2008.
3. Through radiological assessment, subjects with a lymph node length ≥ 10 cm require prior approval from the sponsor before enrollment.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0 -1.
5. QTcF interval ≤450ms in males, and ≤470ms in females.
6. Adequate bone marrow function independent of growth factor and transfusion.
7. Adequate renal and liver function.
8. Willingness by males, female patients of child bearing potential, and their partners to use contraception by effective methods throughout the treatment period and for at least three months following the last dose of study drug.
9. Pregnancy test results of serum samples obtained within 14 days before the first study drug administration in fertile female subjects were negative; If the serum pregnancy test results obtained are> 7 days from the first administration, urine sample obtained before the first study dose of study drug must be negative.
10. Male subjects must avoid sperm donation throughout the treatment period and for at least three months following the last dose of study drug.
11. Ability to understand and willingness to sign a written informed consent form approved by EC committee (the consent form must be signed by the patient prior to any screening or study-specific procedures).
12. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Prior history of allogeneic hematopoietic stem cell transplantation, adoptive cell immunotherapy within 24 months or autologous hematopoietic stem cell transplantation within 12 months.
2. Monoclonal antibody therapy against CLL was adopted within 4 weeks prior to the first dose of the study drug.
3. Receive any of the following treatments within 14 days or 5x half-life before the first dose of study drug, or clinically significant adverse reactions / toxicities due to previous treatments have not recovered to ≤ Grade 1: Anti-tumor therapies include chemotherapy, radiotherapy, anti-tumor steroid treatment, anti-tumor Chinese medicine treatment; investigational treatment, including targeted small molecule drugs.
4. Use the following drugs within 14 days before the first dose of study drug: moderately potent CYP3A inhibitors such as fluconazole, ketoconazole and clarithromycin; moderately potent CYP3A inducers such as rifampin, carbamazepine, phenytoin And St. John's wort.
5. Failure to recover adequately, at the discretion of the investigator, from prior surgical procedures. Patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry.
6. Received Bcl-2 inhibitor treatment.
7. Invasive NHL transformation or central nervous system (CNS) involvement. has occurred.
8. Cardiovascular disease of grade ≥2 (New York Heart Association Class).
9. A significant history of renal, neurological, psychiatric, pulmonary, endocrine, metabolic, immune, cardiovascular or liver disease. The investigator believes that participating in this study will have an adverse effect on him / her. For subjects requiring intervention for any of the above diseases in the past 6 months, the investigator and the sponsor must discuss.
10. Warfarin or other anticoagulants is required.
11. Known to be allergic to study drug ingredients or their analogues.
12. Pregnancy or lactation, or pregnancy is expected during the study period or within 3 months after the last administration of treatment.
13. Within 3 years before entering the study, the subject had a history of active malignant tumors other than CLL / SLL, except that:

    * Fully treated cervical carcinoma in situ;
    * Completely resected basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
    * confinement and resection of previously cured malignancies (or other treatment).
14. Has malabsorption syndrome or other conditions that are not suitable for enteral administration.
15. Uncontrolled other clinically significant symptoms, including but not limited to: uncontrolled systemic infections (viruses, bacteria, or fungi), including but not limited to known hepatitis B virus (HBV) surface antigens and DNA positive(HBV-DNA≥2000copies/mL or ≥500IU/mL); Hepatitis C virus (HCV) antibody positive or RNA positive; human immunodeficiency virus (HIV) antibody positive; Febrile neutropenia occured within 1 week before administration.
16. Primary active autoimmune diseases and connective tissue diseases, such as active and uncontrolled primary autoimmune hemocytopenia, including autoimmune hemolytic anemia (AIHA) and primary immune thrombocytopenia (ITP).
17. Any other condition or circumstance that would, at the discretion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events of APG-2575 single agent | Up to 6 cycles (each cycle is 28 days).
  Adverse events (AE) and serious adverse events (SAE) will be graded according to NCI CTCAE Version 5.0.
Objective Response Rate (ORR) of APG-2575 single agent | Up to 6 cycles (each cycle is 28 days).
  ORR is defined by CR+ CRi + PR(according to NCI-WG CLL(2008)) and by CR+PR ( according to NHL Cheson (2007)).Response will be evaluated every 2 cycles (8 weeks) till complete 6 cycles treatment or one month after last dose.
Dose Limiting Toxicities (DLT) of combination therapy | 28 days.
  DLT will be graded according to NCI CTCAE Version 5.0. DLT will be defined as clinically significant drug-related adverse events during the cycle one.
Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose(RP2D) | 28 days.
  MTD/RP2D will be determined based on DLTs observed during cycle one.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 days.
  Cmax of APG-2575 will be assessed in the patients in single agent or combo study. Cmax of ibrutinib will be assessed in the patients treated with APG-2575 combination with ibrutinib.
Area under the plasma concentration versus time curve (AUC) | 28 days.
  AUC of APG-2575 will be assessed in the patients in single agent or combo study. AUC of ibrutinib will be assessed in the patients treated with APG-2575 combination with ibrutinib.
Objective Response Rate (ORR) of APG-2575 combination therapy | Up to 6 cycles (each cycle is 28 days).
  ORR is defined by CR+ CRi + PR(according to NCI-WG CLL(2008)) and by CR+PR ( according to NHL Cheson (2007)).Response will be evaluated every 2 cycles (8 weeks) till complete 6 cycles treatment or one month after last dose.
Minimal residual lesions (MRD) of peripheral blood and/or bone marrow. | 2 years.
Survival benefit (PFS) of APG-2575 combination therapy | 2 years.
  PFS,Time from the beginning of treatment to the first occurrence of Progressive Disease (PD) or death.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, M.D., Ph.D., Study Director — yzhai@ascentage.com
Locations (18):
- China (18):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial Oncology Hospital, Zhenzhou, Henan
  - Union Hospital medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First affiliated hospital of Soochow University, Suzhou, Jiangsu
  - The First affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Bethune Hospital of Jilin University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang